CLINICAL TRIAL: NCT00818779
Title: Effects of Direct Renin Inhibition on Atherosclerotic Biomarkers in Patients With Stable Coronary Heart Disease and Type 2 Diabetes Mellitus
Brief Title: Direct Renin Inhibition Effects on Atherosclerotic Biomarkers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Tekturna 1
Record Dates: First submitted 2009-01-06; First posted 2009-01-08 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Coronary Artery Disease; Type 2 Diabetes Mellitus
Keywords: diabetes; heart disease; atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2; Diabetes Mellitus; Heart Diseases; Atherosclerosis | interventions — aliskiren; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aliskiren (Experimental): Aliskiren 150-300 mg once daily
  Interventions: Drug: Aliskiren
- Amlodipine (Active Comparator): 5-10 mg amlodipine once daily
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Aliskiren — 150 - 300 mg once daily for 6 weeks
  Other Names: Tekturna
  Arms: Aliskiren
Drug: Amlodipine — 5-10 mg once daily for 6 weeks
  Other Names: Norvasc
  Arms: Amlodipine

SUMMARY:
The investigators aim to assess if a new blood pressure medication, aliskiren, reduces various biomarkers of heart disease found in the blood in patients with a history of both heart disease and type 2 diabetes. The primary hypothesis is that aliskiren will reduce these biomarkers compared to a calcium channel blocker.

DETAILED DESCRIPTION:
Agents that attenuate the renin angiotensin system (RAS), i.e. angiotensin converting enzyme inhibitors (ACE-Is) and angiotensin receptor blockers (ARB), have shown to have therapeutic benefit in a variety of cardiovascular disorders. ACE-Is are considered standard of care for secondary prevention of CAD by the AHA/ACC. Based on the HOPE study, the beneficial effects of ACE-Is in patients at high risk for cardiovascular outcomes may be beyond mere blood pressure control. In addition to their effects on blood pressure, aldosterone, and sodium and water absorption, blockade of the RAS with ACE-Is or ARBs alter key biomarkers of vascular inflammation, vascular endothelial function, and fibrinolytic balance. These surrogate biomarkers are thought to play a role in the progression of atherosclerosis. Biomarkers of vascular inflammation include vascular and intracellular cell adhesion molecule (VCAM and ICAM respectively) and c-reactive protein (CRP). Markers of endothelial function include endothelin-1 (ET-1) and the vasodilator nitric oxide (NO). Plasminogen activator inhibitor-1 (PAI-1) is a prothrombotic marker associated with plaque proliferation and atherosclerosis progression.

ACE-Is block the conversion of angiotensin 1 (Ang 1) to angiotensin 2 (Ang 2). "ACE escape" may attenuate the influence of ACE-Is despite proven benefits in clinical trials.

Aliskiren is the first direct renin inhibitor approved by the FDA for the treatment of hypertension. It is a very specific and potent inhibitor of human renin. As such it may offer an advantage over ACE-I and ARB therapy as it blocks the rate limiting step of the RAS. It does not show a compensatory increase in RAS activity noted with ARBs or non-ACE production of Ang 2 as seen with ACE-Is. Aliskiren appears to have additive blood pressure lowering effects when added to ACE-I or ARB therapy.

A very commonly prescribed antihypertensive, the dihydropyridine calcium channel blocker amlodipine, has a synergistic effect on lowering BP when used with an ACE-I. It has been shown to have mixed effects on atherosclerotic biomarkers in a variety of subjects. Type 2 diabetes affects many of the atherosclerotic markers described above and as such can be a confounding variable in research involving these biomarkers.

With the addition of a new therapeutic agent that affects the RAS, its different pharmacodynamic effects on the RAS compared to ACE-I and ARB therapy, and that Ang 2 levels are not fully blocked by ACE-I therapy, it is critical to better understand how the new class of direct renin inhibitors may influence atherosclerotic biomarkers in patients with a variety of cardiovascular disorders. The objectives of this application are to determine whether the direct renin inhibitor, aliskiren, affects atherosclerotic biomarkers in patients with stable coronary artery disease and diabetes currently receiving standard ACE-I therapy and if aliskiren has a more favorable effect on these markers compared to the calcium antagonist amlodipine.

Large clinical trials have proven the benefit of RAS blockade in reducing cardiovascular morbidity and mortality. The significance of this research is that more information is needed to better understand how antihypertensive agents, particularly those that block the RAS, reduce cardiovascular disease beyond blood pressure reduction alone. Research that elucidates how agents may reduce atherosclerosis is very important to help better target drug therapy to a condition that is the leading cause of death in this country.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* Diagnosis of coronary artery disease
* Currently receiving therapy with an ACE-Inhibitor or Angiotensin Receptor Blocker
* Currently receiving antiplatelet therapy and statin therapy
* Baseline blood pressure > 100/75 mm Hg
* BMI 25-35 kg/m2

Exclusion Criteria:

* Concurrent calcium channel blocker therapy
* Documented peripheral edema
* Hyperkalemia
* Serum creatinine > 2.0
* Diagnosed with proteinuria
* Diagnosed with liver dysfunction or serious rheumatological disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary E Meyerrrose, MD, Principal Investigator — Texas Tech Health Sciences Center Department of Internal Medicine; Brian K Irons, PharmD, Study Director — Texas Tech University Health Sciences Center School of Pharmacy
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aliskiren | Amlodipine
Started | 22 | 16
Completed | 16 | 15
Not Completed | 6 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Amlodipine | Total
Number analyzed (Participants) | 22 | 16 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 15 | 10 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (10) | 63 (16) | 65 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 14 | 10 | 24
Region of Enrollment [Number; unit: participants]
  United States | 22 | 16 | 38

OUTCOME MEASURES:

1. Primary Outcome: Plasminogen Activator Inhibitor 1
Description: Plasminogen Activator Inhibitor 1 is a biomarker found in serum that indirectly assesses blood clotting activity. Lower PAI-1 levels are thought to be better than higher levels. The primary outcome is mean change from baseline and can include negative numbers as a result.
Time Frame: 6 weeks (change from baseline)
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Aliskiren | Amlodipine
Number analyzed (Participants) | 16 | 15
ng/ml | 0.65 [-7.33 to 8.62] | 3.82 [-5.16 to 12.81]

2. Secondary Outcome: Serum Level of Vascular Cell Adhesion Molecule
Description: Surrogate biomarker cardiovascular risk
Time Frame: 6 week (change from baseline)
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Aliskiren | Amlodipine
Number analyzed (Participants) | 16 | 15
ng/ml | -2.4 [-41.1 to 36.3] | -45.9 [-112.8 to 21.0]

3. Secondary Outcome: Serum Level of Intracellular Cell Adhesion Molecule
Description: Surrogate biomarker of cardiovascular risk
Time Frame: 6 week (change from baseline)
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Aliskiren | Amlodipine
Number analyzed (Participants) | 16 | 15
ng/ml | -4.9 [-17.2 to 7.4] | -10.3 [-31.2 to 10.6]

4. Secondary Outcome: Serum Level of C-reactive Protein
Description: Surrogate biomarker of cardiovascular risk
Time Frame: 6 week (change from baseline)
Measure: Mean (95% Confidence Interval); unit: mg/l
Arm/Group | Aliskiren | Amlodipine
Number analyzed (Participants) | 16 | 15
mg/l | 0.0397 [-0.2310 to 0.3104] | 0.1032 [-0.1974 to 0.4038]

5. Secondary Outcome: Serum Level of Nitric Oxide
Description: Surrogate biomarker of cardiovascular risk
Time Frame: 6 week (change from baseline)
Measure: Mean (95% Confidence Interval); unit: mmmol/l
Arm/Group | Aliskiren | Amlodipine
Number analyzed (Participants) | 16 | 15
mmmol/l | 2.66 [-7.45 to 12.76] | 7.49 [-1.43 to 16.41]

ADVERSE EVENTS:
Arm/Group | Aliskiren | Amlodipine
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/22 | 0/16

LIMITATIONS AND CAVEATS:
Small sample size led to large standard deviation in biomarkers assessed and limited power to detect a diffference

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes